CLINICAL TRIAL: NCT03432325
Title: Neural Enabled Prosthesis for Upper Limb Amputees
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ranu Jung, Executive Director and Endowed Chair for I3R, Distinguished Professor, Associate Vice Chancellor, University of Arkansas, Fayetteville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NEP601; R01EB023261 (NIH); CDMRP-E00915.1a (Other: Human Research Protection Office); W81XWH1910839 (Other Grant/Funding Number: USAMRAA)
Record Dates: First submitted 2018-01-05; First posted 2018-02-14 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Amputation Arm and Hand, Unilateral Right; Amputation Arm and Hand, Unilateral Left; Prosthesis User

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Neural Enabled Prosthesis (Experimental): Neural Enabled Prosthesis Treatment Group
  Interventions: Device: Neural Enabled Prosthesis

INTERVENTIONS:
Device: Neural Enabled Prosthesis — Surgically implanted neural enabled prosthesis

SUMMARY:
This study is designed to evaluate the feasibility of The Adaptive Neural Systems Neural-Enabled Prosthetic Hand (ANS-NEPH) system.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a new prosthetic system for transradial amputees called the neural-enabled prosthetic hand (ANS-NEPH). It is intended to provide the sense of touch, grasp force and hand opening to the user by sending electrical stimulation pulses to electrodes implanted in nerve fascicles in the upper arm of the residual limb. The system uses measurements from sensors in the prosthetic hand and wireless communication to the implanted neurostimulator to adjust the pulses continuously so that the user gets sensation as tasks are performed with the prosthesis.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral transradial amputation
2. Amputation occurred 9 months ago or more
3. Functional hand contralateral to the amputation
4. Ability and willingness to use myoelectric arm (as determined by prosthetist)
5. 18 years of age or older
6. Ability to obtain transportation to the research site and the clinicians' offices
7. U.S. citizen or permanent U.S. resident
8. Signed the Informed Consent Form

Exclusion Criteria:

1. Absence of limb due to birth defect
2. Evidence of denervation of the residual limb
3. Phantom limb pain that is severe enough to impair or restrict activity
4. Any neurological condition affecting motor and/or sensory function that would interfere with use of the intact hand or residual limb (as determined by neurologist)
5. Visual impairment that would affect hand usage during experimental procedures
6. History of chronic infections
7. History of recurring ulcers or blisters on the residual limb
8. Evidence of an active infection, non-healed ulcer, recent history of a healed ulcer (< 3 months)
9. Use of another implanted electrical device (such as a pacemaker or nerve stimulator)
10. Undergoing diathermy therapy of the residual limb
11. History of non-compliance with medical or research procedures or any condition that would limit their ability to comply with study related procedures (self-reported)
12. Self-reported emotional or psychological disorders or history of drug or alcohol abuse or addiction
13. Memory disorders or significant cognitive impairment (self-reported and/or clinical observation during consent and screening procedures)
14. Moderate to severe chronic pain
15. Pregnant or nursing
16. Self-reported sensitivity to material derived from porcine source
17. Enrolled in another investigational research study
18. Any medical or psychiatric condition not otherwise specified (such as uncontrolled high blood pressure, heart or lung disease, active infection, and serious metabolic disorders) that would expose the subject to unacceptable risk and/or limit their ability to perceive meaningful sensation from stimulation of the peripheral nerves of the residual limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of the Neural Stimulation System | Up to 104 weeks - post-treatment
  Documented as the number of treatment-related adverse events as assessed by CTCAE v4.0.

SECONDARY OUTCOMES:
Efficacy: Functionality of implanted system components | Up to 104 weeks - post-treatment
  Documented as the percentage of implanted electronic units fully operational and the percentage of electrodes intact (having measured impedance values < OR = 30kΩ)
Efficacy: Elicited sensations | Up to 104 weeks - post-treatment
  Ability of the system to elicit graded sensations documented as the correlation between stimulation intensity (expressed as a percentage of the stimulation range) and reported intensity of the elicited sensation (expressed as a percentage of the range of elicited sensations)
Efficacy: Graded control | Up to 104 weeks - post-treatment
  The ability of the system to enable graded control of a prosthesis measured as the accuracy with which the subject can achieve a specified target level of grasp force or hand opening. Comparing performance with & without sensory stimulation
Efficacy: Activity Measure for Upper Limb Amputees (AM-ULA) | Baseline plus up to 104 weeks post-treatment
  The ability of the system to facilitate completion of functional tasks documented by using the AM-ULA. Comparing performance with & without sensory stimulation
Clinical Surveys: Orthotics and Prosthetics User Survey - The Upper Extremity Functional Status (OPUS - UEFS) | Baseline plus up to 104 weeks post-treatment
  The UEFS is a 28-item self-report pertaining to an individual's performance of self-care and daily living skills using the prosthetic hand. UEFS has a 5-point Likert scale where Score Points are 0 = not able, 1 = difficult, 2 = easy, 3 = very easy scores are given. The survey will be used to document changes in participants' functional status and quality of life.
Clinical Surveys: Disabilities of the Arm, Shoulder, and Hand (DASH) | Baseline plus up to 104 weeks post-treatment
  The DASH Outcome Measure is a 30-item (scored 1-5) self-report questionnaire designed to measure physical function and symptoms in people with any of several musculoskeletal disorders of the upper limb. The survey will be used to measure disability of the upper extremities, and monitor change or function over time.
Clinical Surveys: Trinity Amputation and Prosthetics Experience Scales - Revised (TAPES-R) | Baseline plus up to 104 weeks post-treatment
  This outcome measure is a 54-item self-report, health-related QOL questionnaire. This survey will be used to measure psychosocial processes that are linked with adapting to a prosthesis, to the activity restrictions associated with wearing a prosthesis, and to satisfaction with the prosthesis. Only some sections of the complete version have been included in the survey documents. In specific, we will administer the Psychosocial Scale (15 items) and Satisfaction with the Prosthesis Scale (8 items).
Clinical Surveys: Groningen Questionnaire - Problems After Arm Amputation (GQ-PAAA) | Baseline plus up to 104 weeks post-treatment
  The GQ_PAAA is a 14-item self-report measurement. This survey will be used to document frequency of phantom limb sensation, phantom limb pain, and stump pain. A modified version of this measure has been included in the survey documents.
Clinical Surveys: 12-Item Short Form Survey (SF-12) | Baseline plus up to 104 weeks post-treatment
  This outcome measure is a 12-item self-report questionnaire that provides glimpses into mental and physical functioning and overall health-related-quality of life. This survey will be used to document health-related quality of life.
Clinical Surveys: McGill Pain Questionnaire (MPQ) | Baseline plus up to 104 weeks post-treatment
  This survey will be used to document the quality and intensity of pain that the participant is experiencing. Participants select a single word from each of the 20 groups and then describe their present pain intensity on a scale of 0 to 5.
Clinical Assessment: Adaptive Neural Systems - Phantom Limb Telescoping Assessment (ANS-PLTA) | Baseline plus up to 104 weeks post-treatment
  We have developed this assessment to measure the phantom limb telescoping at the beginning and at the end of each session to track how the length of the phantom limb changes after stimulation within a session and across sessions as reported by the subject. Subjects report where the end of the phantom limb is by pointing at it with the other hand.
Clinical Assessment: The Southampton Hand Assessment Procedure (SHAP) | Baseline plus up to 104 weeks post-treatment
  SHAP is a clinically validated hand function test developed to assess the effectiveness of upper limb prostheses. The SHAP is made up of 6 abstract objects and 14 Activities of Daily Living (ADL). Each task is timed by the subject and recorded on an assessment sheet by the assessor.

CONTACTS AND LOCATIONS:
Overall Officials: Ranu Jung, Ph.D., Principal Investigator — University of Arkansas, Fayetteville; Paul Pasquina, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (2):
- United States (2):
  - University of Arkansas, Fayetteville, Arkansas
  - Walter Reed National Military Medical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No
The study is a feasibility study therefore data collected is being used to assess the feasibility of the system for future investigation.